CLINICAL TRIAL: NCT05231486
Title: Effectiveness of the Cognitive Orientation to Daily Occupational Performance Group Approach for Children With Developmental Coordination Disorder (DCD) - ECOOPG
Brief Title: Effectiveness of the COOP Group Approach for Children With Developmental Coordination Disorder (DCD)
Acronym: ECOOPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université du Québec à Trois-Rivières (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL20_0429
Record Dates: First submitted 2021-12-28; First posted 2022-02-09 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Developmental Coordination Disorder
Keywords: Cognitive Orientation to daily Occupational Performance (CO-OP); Single Case Experimental Design (SCED); Developmental Coordination Disorder (DCD); Group intervention
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Intervention Model Description: The study design is similar to a matched case-control study using Single Case Experimental Design (SCED) methodology with a multiple baseline design across subjects.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cognitive Orientation to daily Occupational Performance 1 (Experimental): This arm is the first group composed of four childrens who will do the CO-OP. CO-OP uses cognitive problem solving techniques to facilitate motor skill acquisition. The therapist facilitates with guided discovery the child to generate solution for problems in their performance areas.
  The four patients will begin the sessions one week apart each.
  Interventions: Behavioral: Cognitive Orientation to daily Occupational Performance
- Cognitive Orientation to daily Occupational Performance 2 (Experimental): This arm is the second group composed of four others childrens who will do the CO-OP.
  CO-OP uses cognitive problem solving techniques to facilitate motor skill acquisition. The therapist facilitates with guided discovery the child to generate solution for problems in their performance areas The four patients will begin the sessions one week apart each.
  Interventions: Behavioral: Cognitive Orientation to daily Occupational Performance
- Cognitive Orientation to daily Occupational Performance 3 (Experimental): This arm is the third group composed of four others childrens who will do the CO-OP.
  CO-OP uses cognitive problem solving techniques to facilitate motor skill acquisition. The therapist facilitates with guided discovery the child to generate solution for problems in their performance areas The four patients will begin the sessions one week apart each.
  Interventions: Behavioral: Cognitive Orientation to daily Occupational Performance
- Cognitive Orientation to daily Occupational Performance 4 (Experimental): This arm is the fourth group composed of four others childrens who will do the CO-OP.
  CO-OP uses cognitive problem solving techniques to facilitate motor skill acquisition. The therapist facilitates with guided discovery the child to generate solution for problems in their performance areas The four patients will begin the sessions one week apart each.
  Interventions: Behavioral: Cognitive Orientation to daily Occupational Performance
- Cognitive Orientation to daily Occupational Performance 5 (Experimental): This arm is the fifth group composed of four others childrens who will do the CO-OP.
  CO-OP uses cognitive problem solving techniques to facilitate motor skill acquisition. The therapist facilitates with guided discovery the child to generate solution for problems in their performance areas The four patients will begin the sessions one week apart each.
  Interventions: Behavioral: Cognitive Orientation to daily Occupational Performance

INTERVENTIONS:
Behavioral: Cognitive Orientation to daily Occupational Performance — CO-OP uses cognitive problem solving techniques to facilitate motor skill acquisition. The therapist facilitates with guided discovery the child to generate solution for problems in their performance areas.

SUMMARY:
Developmental Coordination Disorder (DCD) is a neurodevelopmental disorder that causes difficulty in motor coordination both in their learning and in their execution. This disorder affects about 5% of school-age children. The Cognitive Orientation to daily Occupational Performance (CO-OP) approach is a non-drug intervention technique, focused on solving motor problems where the patient is taught cognitive strategies (in small groups) with a view to acquire and execute motor coordination effectively. It is part of Cognitive-Behavioral techniques (CBT). This is one of the approaches recommended internationally and in France for patients with Developmental Coordination Disorder. In addition, for DCD patients, non-drug interventions in small groups are recommended internationally for this condition. However, few studies are available to validate the CO-OP approach in this format. Since 2013, the Department of Child and Adolescent Psychological Medicine sector 2 (MPEA2) of the University Hospital of Montpellier has offered group interventions for children diagnosed with DCD who are referred to them in current care practice with the CO-OP approach. In view of the major repercussions of DCD on self-esteem, academic and academic success and the development of social ties, this group therapy will restore a life trajectory and improve the quality of life of these patients.

DETAILED DESCRIPTION:
Methodology:

The study design used is Single Case Experimental Design (SCED) methodology with multiple baseline design across subjects. The principle of SCED is based on the fact that each subject is his own control. The judgment criterion is repeated at least 5 times before initiating the intervention (Baseline phase), then repeated during the intervention (intervention phase) and after intervention (follow-up phase). It is the demonstration of 3 effects, represented here by at least 3 patients in parallel per group, which leads to the conclusion that the intervention is effective.

The children will be randomly integrated into the protocol according to the Wampold - Worsham procedure. Each child will be randomly assigned to the 4 potential positions, shifted in the multiple baseline plane of the SCED protocol of this study.

The SCED methodology uses an analysis of data and statistics specifics. The first phase of analysis will be a visual analysis of the differential between two contiguous phases on three specific aspects: the level, the trend and the variability of the dependent variable studied. Then, a statistical analysis specific to SCED protocols is possible. The use of random sequential introduction procedure such as Wampold - Worsham allows to extract a p value for each patient. This probability p is based on the rank of the mean corresponding to the real transitions among other hypothetical possible transitions of the SCED protocol. Then, the statistical analysis takes into account the overlap rate by calculating the number of overlapping points between the phases : the more overlap there is between two phases, the less the intervention effect is present. Conversely, if two phases show no overlap of measures, the intervention is likely to have a larger effect. Many overlap techniques exist. Those used for this study will be the "Non-overlap of All Pairs - NAP" technique, the Tau-U and Tau-U corrected from the baseline.

The main dependent variable is an evaluation of the performance level of target motor coordination worked for each patient in groups on video with the Performance Quality Rating Scales (PQRS). The PQRS is a 10-point Likert scale used to assess performance and change in performance directly during the patient's motor performance recorded on video for this study. The PQRS is a Likert scale from 1 (very poor performance) to 10 (very strong performance) conventionally used in the literature on CO-OP. The performance criteria will be determined for each point of the Likert scale a priori for each objective.

Two independent assessors trained in CO-OP and PQRS will assess children's motor performance, once all the videos have been collected, anonymized and randomized as to their temporal place in the protocol. The motor performance of each child on each task will be evaluated from a minimum of 5 video recordings for each phase of the protocol (Baseline, Intervention, Follow-up). For the total duration of the study, a sample of a minimum of 20 records and a maximum of 23 records per target task, for each child will be used. The videos will be produced each week of the protocol within the Montpellier University Hospital.

Additionally, a computerized spontaneous tapping task of about one minute will be offered at the end of each session in order to measure the average frequency and the variability.

Finally, the KIDSCREEN-27 questionnaire will be used. This tool subjectively assesses the health and well-being of children and adolescents (health-related quality of life, HRQH). Two questionnaires (child and proxy version) will be completed during the first session and during the last session at the Montpellier University Hospital.

Number of patients:

It is planned to include 20 patients. Five groups comprising four patients will be proposed.

SCED studies must provide proof of efficacy by replicating the effects on at least 3 patients within a single publication. However, international recommendations indicate that proof of the effect requires 20 combined cases in order to demonstrate the proof of effectiveness of an intervention with this type of design.

Patient selection: from wait-list for CO-OP intervention in MPEA2 unity of University Hospital Center (CHU) of Montpellier

Duration of project: 36 month Inclusion period: 36 month Duration of experimental procedure : 23 week (approximately 6 month) Duration of statistical analyzes / valuation: 6 months Estimated duration of the study: 48 months (from M0 to M48)

Schedule visit: 23 sessions maximum per patient

Phase A - Sessions 1 to 8 - baseline :

A first telephone contact is made in order to propose entry into the family study. Once the 4 inclusions per group have been made, a draw is made to determine the family's inclusion session. An individual interview on entering the study will be carried out and will last for one hour. This interview allows on the one hand to explain the CO-OP approach and on the other hand to determine the specific objectives defined by the patient and his family. For this, the semi-structured interview using the Canadian Occupational Performance Measure will be carried out. This interview is performed for each child before their inclusion in the study. During this interview, the first KIDSCREEN-27 questionnaire (child version and proxy version (parent)) is completed by the child and his parents

A first meeting including all the families and children of a group (4 families) participating in the study will be offered just before session 1 (start of phase A - Baseline). This meeting will last thirty minutes and will be devoted to explaining the course of the following sessions (sessions 2 to 8, phase A) as well as the selection of 3 target activities that will be worked on during the CO-OP intervention among the 5 initially selected. The 2 activities not worked on during the protocol will allow a measurement of the transfer effects of the CO-OP intervention.

In session 1, one child (randomly selected, child 1) begins the individual baseline control phase (A) and continues until the 8th session, while children 2 to 4 remain out of the baseline condition. A. The inclusion procedure (phase A) begins for another child (randomly selected, child 2) from session 2 and continues for child 2 until the 8th session, while children 3 and 4 remain outside phase A. Finally, the last children (chosen at random, children 3 and 4) enter their phase A in the same way from sessions 3 for the child 3 and session 4 for the child 4. This phase is the randomized individual inclusion phase (4). Phase A (Baseline) ends after the 8th session.

Overall child 1 will have 23 sessions, child 2 will have 22 sessions, child 3 will have 21 sessions and child 4 will have 20 sessions.

Families will have three options in order to take the necessary measures during the pre-intervention phase (phase A, Baseline, session 1 to 8):

* Come to the CHU
* Make a ZOOM videoconference and record the motor performances necessary for the family home (PQRS and Motrice task (tapping))
* Offer a reminder phone call from the therapists to take the measurements at the family home From session 4, all inclusions of a group (4 participants) will be made for the Baseline phase.

During the rest of phase A (session 4 to 8), the children will have to carry out the 5 motor activities, without intervention of the therapists in order to assess the maintenance of the target motor coordination targets worked and to carry out the control measurement (spontaneous tapping, measurement of frequency and variability).

The same will the same for the other 16 children to be included in the study. The selection will be made in groups for 4 children.

Phase B - Sessions 9 to 18 - Intervention :

Phase B (intervention) begins in session 9 with the CO-OP approach. The sessions will be filmed in full from sessions 9 to 18. The procedural fidelity, that is to say the respect of the active principles of the CO-OP by the therapists, will be measured from three sessions filmed in full and chosen from randomly among the 10 that will be carried out (30%) during the intervention phase (session 9 to 18).

A Phase B - Intervention exit meeting with all families and children will be offered immediately after session 18.

Phase C - Sessions 19 to 23 - post-intervention :

Finally, from session 19 to 23 (post-intervention, Follow-up, phase C), families will have the same possibilities as phase A in order to take the necessary measures on post-intervention phase C (Follow-up, session 19 to 23 ).

During the rest of the Follow-up (session 19 to 23), as for phase A (session 4 to 8), the children will have to carry out the 5 motor activities, without intervention of the therapists in order to assess the maintenance of the target motor coordination targets worked on and perform control measurement (spontaneous tapping, frequency and variability measurement). Non-motor group games will be performed the rest of the time.

Concerning the individual exit interview, child 1 will carry out this interview in session 20, child 2 in session 21 and child 3 in session 22 and child 4 in session 23. These interviews will be carried out in parallel with the sessions included in the follow-up phase and consists of performing the Canadian Occupational Performance Mesure (COPM).

During session 23, which must be carried out face-to-face, children and parents must again complete the KIDSCREEN-27 questionnaires (patient and proxy version) at the end of the protocol, in addition to carrying out the 5 motor activities, without intervention from the therapists. and perform the control measurement (spontaneous tapping).

The rhythm of the sessions is 1 session per week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DCD formally established during a multidisciplinary assessment, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria
* 8-12 years
* Present in wait list for CO-OP intervention
* Parents consent

Exclusion Criteria:

* Language disorder
* High level of anxious
* Low level of motivation
* Participation to another intervention
* Subject refusal to participate
* Parental refusal to participate

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Performance Quality Rating Scale (PQRS) | Up to 23 weeks
  The performance quality rating scale (PQRS) is an observational, video-based tool intended to measure the actual performance of individual client-selected activities.
  The PQRS is a Likert scale from 1 (very low performance) to 10 (very high performance) classically used in the literature on CO-OP.

SECONDARY OUTCOMES:
Free tapping | Up to 23 weeks
  Tasks of free tapping are used to assess motor timing. Free tapping is a validated experimental paradigm to investigate the speed and consistency of self-produced finger tapping and has been used wi[h adults and childrens. The subjects were required to tap a response button with the right finger 80 times as regularly as possible at a freely chosen rhythm. The reaction times reflect the preferred speed, while the consistency and regularity of the motor production is reflected by the variability of response.
KIDSCREEN-27 | Up to 23 weeks
  The KIDSCREEN-27 Questionnaires assess children's and adolescents' subjective health and well-being (health-related quality of life, HRQOL). the KIDSCREEN assesses HRQOL in Physical and Psychological Well-Being (12 items), Autonomy & Parents (7 items), Peers & Social Support (4 items), and School Environment (4 items).It was developed as a self-report measure applicable for healthy and chronically ill children and adolescents aged from 8 to 18 years.

CONTACTS AND LOCATIONS:
Overall Officials: Amaria BAGHDADLI, Principal Investigator — MPEA2, Département Universitaire de Pédopsychiatrie, CHU de Montpellier
Locations (1):
- Hôpital de la Colombière (CHU), Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Data will be made available to persons who address a reasonable dataset request to the principal investigator (c/o Emmanuel Madieu).
  In accordance with current regulations in France, the data may be made available after obtaining approvals from regulatory bodies (CPP, CESREES, CNIL, etc.). In accordance with GDPR, participants must be individually informed of the sharing of their data. The data will then be available via Nextcloud CHU tools. The data can then be used for all analyses.
Supporting Information: Study Protocol
Time Frame: Datasets can be requested 24 month after the end of the study.
  The protocol will be made available after publication in scientific journal.
Access Criteria: The conditions under which members of the public will be granted access to datasets are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
  * The appropriate CNIL approval has been obtained by the user.

REFERENCES:
- [Derived] Madieu E, Therriault PY, Cantin N, Baghdadli A. Effectiveness of CO-OP group intervention for children with developmental coordination disorder: single-case experimental design study protocol. BMJ Open. 2023 Dec 30;13(12):e073854. doi: 10.1136/bmjopen-2023-073854. PMID 38159958